CLINICAL TRIAL: NCT06279195
Title: Comprehensive Mechanistic Phenotyping of Idiopathic Pelvic Pain With Real-time Uterine Imaging and Relugolix-Combination Therapy Treatment
Brief Title: Phenotyping of Idiopathic Pelvic Pain With Real-time Uterine Imaging and Relugolix-Combination Therapy Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not obtain approval for the planned study with available funding
Sponsor: Endeavor Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Kevin Hellman, Research Associate Professor, Endeavor Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EH23-326
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Pain
Keywords: Idiopathic Pelvic Pain; Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — relugolix; Estradiol; Norethindrone Acetate; Tablets

STUDY DESIGN:
Intervention Model Description: Participants in two groups with different conditions will be give REL-CT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Idiopathic Pelvic Pain (Experimental): Participants with Idiopathic Pelvic Pain must: 1. Self-report an average non-menstrual pelvic pain rating of ≥ 4/10 (on a 0 to 10 Numeric Rating Scale) over the past 6 months. 2. Not have received a prior diagnosis attributed to a secondary cause (e.g., leiomyoma, endometriosis). Participants will be instructed to start taking Relugolix-combination therapy (40 mg of relugolix, 1 mg of estradiol, and 0.5 mg of norethindrone acetate) within 7 days of their period starting, at the same time every day for the next 6 months.
  Interventions: Drug: Relugolix (40 mg) /estradiol (1 mg)/norethisterone acetate (0.5 mg) oral tablet
- Endometriosis: (Experimental): Participants with Endometriosis: 1. Must self-report an average non-menstrual pelvic pain rating of ≥ 4/10 (on a 0 to 10 Numeric Rating Scale) over the past 6 months. 2. Have a previously confirmed surgical diagnosis of stage III-IV endometriosis, indicating potential remission. Participants will be instructed to start taking Relugolix-combination therapy (40 mg of relugolix, 1 mg of estradiol, and 0.5 mg of norethindrone acetate) within 7 days of their period starting, at the same time every day for the next 6 months.
  Interventions: Drug: Relugolix (40 mg) /estradiol (1 mg)/norethisterone acetate (0.5 mg) oral tablet

INTERVENTIONS:
Drug: Relugolix (40 mg) /estradiol (1 mg)/norethisterone acetate (0.5 mg) oral tablet — All participants will be instructed to take REL-CT.
  Other Names: Myfembree; Relugolix Combination Therapy; REL-CT

SUMMARY:
The mechanisms underlying variable efficacy of Relugolix-Combination Therapy (REL-CT) in mitigating unexplained pelvic pain will be evaluated with uterine imaging techniques and quantitative sensory testing.

DETAILED DESCRIPTION:
The mechanisms underlying variable efficacy of Relugolix-Combination Therapy (REL-CT) in mitigating unexplained pelvic pain will be evaluated with real-time uterine imaging techniques and quantitative sensory testing. Advanced MRI methodology enables the assessment of various uterine parameters, including contractions, peristalsis, perfusion, blood oxygenation, and structural factors. Importantly, it is possible to temporally correlate these mechanisms with self-reported spontaneous menstrual cramping pain through real-time imaging.

In the first aim of this proposal (Aim #1), mechanisms underlying unexplained menstrual pain phenotypes linked to deficiencies in myometrial activity, perfusion, and oxygenation and evaluate the subsequent impact of REL-CT will be evaluated. Aim #2 focuses on characterizing unexplained menstrual pain phenotypes associated with impairments in the central nervous system sensory functions and the effects of REL-CT. Quantitative sensory testing methods will be used to comprehensively assesses peripheral, central ascending, central integrating, and central descending nervous system components related to pelvic pain. In the past, this testing can identify central nervous system component pain that predicts the pain trajectory and corresponds with treatment outcomes.

By analyzing the relationship between the variable effectiveness of REL-CT treatment to observed mechanisms in menstrual pain, it may possible to identify specific unexplained pelvic pain phenotypes amenable to medical management. Furthermore, because that the precise mechanisms by which REL-CT alleviates menstrual pain in endometriosis remain incompletely understood, a cohort of endometriosis patients will be also studied. The overarching objective is to uncover the underlying mechanisms that advance the comprehension of menstrual pain biology and establish these mechanisms as phenotypic markers for treating REL-CT.

ELIGIBILITY:
Inclusion Criteria

Idiopathic pelvic pain (40 participants):

* Self-report an average non-menstrual pelvic pain rating of ≥ 2/10 (on a 0 to 10 Numeric Rating Scale) over the past 6 months.
* Not have received a prior diagnosis attributed to a secondary cause (e.g., leiomyoma, endometriosis).

Endometriosis (20 participants)

* Self-report an average non-menstrual pelvic pain rating of ≥ 2/10 (on a 0 to 10 Numeric Rating Scale) over the past
* Previously confirmed surgical diagnosis of stage III-IV endometriosis, indicating potential remission.

Exclusion Criteria:

* History of blood clots,
* Allergies to REL-CT ingredients
* Diabetes
* Migraines
* Osteoporosis
* Vascular disease
* Hormone-sensitive cancers
* Smoking.
* Missing limbs
* Paralysis,
* Conditions associated with irregular menses
* Congenital conditions affecting reproductive function
* Intrauterine device use
* Pelvic inflammatory conditions
* Active genitourinary infections,
* Inability to read or comprehend the informed consent document written in English
* History of metallic implants, history of metallic injury, any condition precluding investigation with MRI
* BMI exceeding 40
* Uncontrolled thyroid dysfunction
* Adrenal dysfunction
* Renal disorders
* Liver disorders
* Coagulopathy,
* Gastrointestinal conditions or surgeries that may affect absorption

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between post-treatment pelvic pain and baseline uterine contraction frequency | 6 months
  At baseline before intervention, the number of contractions over a 10 minute period will be measured with MRI.Participants will complete a pain diaries before REL-CT treatment and 6 months after starting REL-CT treatment. Participants will be asked to rate their overall pelvic, bladder test pain and bowel pain at the end of the day via REDCap (on 0-10 scale, 0 no pain, 10 worst pain imaginable). The average pain ratings during non-menstrual days will be used to generate continuous ratings of pelvic pain for each diary. The correlation coefficient between the amount of contractions measured with MRI and average non-menstrual pelvic pain will be calculated.
Correlation between post-treatment pelvic pain and baseline sensory hypersensitivity Z-score. | 6 months
  A composite Z-scored total sensory hypersensitivity score will be calculated by summing the z-scores obtained from the baseline sensory tests during bladder pain, bodily pressure pain threshold, and visual/audio tests at baseline. The correlation coefficient between the Z-scored total sensory hypersensitivity scored and average non-menstrual pelvic pain will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized data with potentially interested experience scientific researchers. Shared data includes pain diary, questionnaire data, MRI data, and sensory testing data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in pelvic pain. Data or samples shared will be coded, with no personally identifying included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.

REFERENCES:
- [Background] Hellman KM, Kuhn CS, Tu FF, Dillane KE, Shlobin NA, Senapati S, Zhou X, Li W, Prasad PV. Cine MRI during spontaneous cramps in women with menstrual pain. Am J Obstet Gynecol. 2018 May;218(5):506.e1-506.e8. doi: 10.1016/j.ajog.2018.01.035. Epub 2018 Feb 2. PMID 29409786
- [Background] Kmiecik MJ, Tu FF, Silton RL, Dillane KE, Roth GE, Harte SE, Hellman KM. Cortical mechanisms of visual hypersensitivity in women at risk for chronic pelvic pain. Pain. 2022 Jun 1;163(6):1035-1048. doi: 10.1097/j.pain.0000000000002469. Epub 2021 Aug 27. PMID 34510138